CLINICAL TRIAL: NCT02798120
Title: A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris
Brief Title: P3 Long Term Safety Study of Once Daily SB204 in Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-AC303
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB204 4% (Experimental): All subjects received SB204 4% once daily (QD) in this open label study. Subjects assigned to SB204 4% QD in the parent study (NI-AC301/302) continued to receive SB204 for 40 more weeks. Subjects assigned to Vehicle Gel in the parent study (NI-AC301/302) received SB204 4% QD in this open label study.
  Interventions: Drug: SB204 4%

INTERVENTIONS:
Drug: SB204 4% — Open label, topical SB204 4%
  Other Names: NVN1000

SUMMARY:
This is a multi-center, open label long-term safety (LTS) study to be conducted in approximately 600 subjects with acne vulgaris.

DETAILED DESCRIPTION:
A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Have completed 12 weeks of treatment in NI-AC301 or NI-AC302

Exclusion Criteria:

* Terminated early from an SB204 Phase 3 pivotal study for any reason
* Have an on-going adverse event at Week 12 visit for NI-AC301 or NI-AC302 that warrants stopping study drug application
* Have used medications or vitamins during the 12 weeks immediately preceding this study which were reported to exacerbate acne.

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, Study Chair — Novan, Inc.
Locations (69):
- United States (69):
  - CIL #138, Birmingham, Alabama
  - CIL #218, Mobile, Alabama
  - CIL #189, Phoenix, Arizona
  - CIL #146, Anaheim, California
  - CIL #139, Cerritos, California
  - CIL #216, Chula Vista, California
  - CIL #186, Fresno, California
  - CIL #210, Fresno, California
  - CIL #174, Huntington Beach, California
  - CIL #213, La Mesa, California
  - CIL #209, Oceanside, California
  - CIL #190, Sacramento, California
  - CIL #161, San Diego, California
  - CIL #113, San Diego, California
  - CIL #195, Santa Ana, California
  - CIL #119, Santa Monica, California
  - CIL #199, Santa Rosa, California
  - CIL #103, Boca Raton, Florida
  - CIL #208, Hialeah, Florida
  - CIL #212, Homestead, Florida
  - CIL #222, Lauderdale Lakes, Florida
  - CIL #170, Miami Lakes, Florida
  - CIL #204, Miami Springs, Florida
  - CIL #172, Orlando, Florida
  - CIL #185, Ormond Beach, Florida
  - CIL #203, Ormond Beach, Florida
  - CIL #110, Pinellas Park, Florida
  - CIL #227, Sanford, Florida
  - CIL #211, South Miami, Florida
  - CIL #176, St. Petersburg, Florida
  - CIL #152, Tampa, Florida
  - CIL #229, Tampa, Florida
  - CIL #144, Tampa, Florida
  - CIL #153, Wellington, Florida
  - CIL #116, Newnan, Georgia
  - CIL #143, Savannah, Georgia
  - CIL #175, New Albany, Indiana
  - CIL #191, Overland Park, Kansas
  - CIL #215, Wichita, Kansas
  - CIL #117, Louisville, Kentucky
  - CIL #194, Richmond, Kentucky
  - CIL #219, Monroe, Louisiana
  - CIL #187, St Louis, Missouri
  - CIL #148, Norfolk, Nebraska
  - CIL #140, Omaha, Nebraska
  - CIL #182, Las Vegas, Nevada
  - CIL #201, Berlin, New Jersey
  - CIL #141, Montclair, New Jersey
  - CIL #156, Albuquerque, New Mexico
  - CIL #108, Rochester, New York
  - CIL #221, Salisbury, North Carolina
  - CIL #169, Cincinnati, Ohio
  - CIL #226, Cincinnati, Ohio
  - CIL #237, Gresham, Oregon
  - CIL #200, Portland, Oregon
  - CIL #137, Broomall, Pennsylvania
  - CIL #178, Philadelphia, Pennsylvania
  - CIL #217, Chattanooga, Tennessee
  - CIL #198, Arlington, Texas
  - CIL #160, Austin, Texas
  - CIL #154, Beaumont, Texas
  - CIL #184, Bryan, Texas
  - CIL #188, Houston, Texas
  - CIL #151, Plano, Texas
  - CIL #168, Plano, Texas
  - CIL #224, San Antonio, Texas
  - CIL #106, Salt Lake City, Utah
  - CIL #105, Lynchburg, Virginia
  - CIL #231, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who successfully completed one of the pivotal parent studies NI-AC301 and NI-AC302 were eligible to roll over into NI-AC303. Those subjects assigned to SB204 once daily (QD) in the parent study continued to receive open label SB204 for 40 more weeks (total ~52 weeks) and are denoted as SB204 experienced. Those subjects assigned to vehicle gel in the parent study were rolled over and received open label SB204 in this trial (total ~40 weeks of SB204 treatment) and are denoted SB204 naive.
Groups:
- SB204 4% Experienced: Subjects who received SB204 4% in the parent study (NI-AC301 or NI-AC302) were considered SB204 experienced at the time of enrollment into NI-AC303.
- SB204 Naive: Subjects who received vehicle gel in the parent study (NI-AC301 or NI-AC302) were considered SB204 naive at the time of enrollment into this study (NI-AC303). They began treatment with SB204 on the day of enrollment.
Period: Overall Study
Arm/Group | SB204 4% Experienced | SB204 Naive
Started | 296 | 305
Completed | 232 | 216
Not Completed | 64 | 89

BASELINE CHARACTERISTICS:
Population: Safety population. As this was an open label, long term safety study, all subjects were in the safety population.
Groups:
- SB204 Experienced: Subjects who were assigned to and received SB204 in the pivotal study (NI-AC301 or NI-AC302) were denoted as being SB204 experienced when they rolled over into the open-label long term safety study (NI-AC303). These subjects were on treatment with SB204 for up to 52 weeks (12 weeks in the pivotal study + 40 weeks in this study.
- SB204 Naive: Subjects who were assigned to and received Vehicle Gel in the pivotal study (NI-AC301 or NI-AC302) were denoted as being SB204 naive when they rolled over into the open-label long term safety study (NI-AC303). These subjects were on treatment with SB204 for up to 40 weeks.
- Total: Total of all reporting groups
Arm/Group | SB204 Experienced | SB204 Naive | Total
Number analyzed (Participants) | 296 | 305 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (8.86) | 21.0 (8.66) | 21.2 (8.76)
Age, Customized [Count of Participants; unit: Participants]
  Juvenile (<18 years) | 133 | 149 | 282
  Adult (≥18 years) | 163 | 156 | 319
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 183 | 357
  Male | 122 | 122 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 122 | 233
  Not Hispanic or Latino | 185 | 183 | 368
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 19 | 42
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 58 | 56 | 114
  White | 211 | 221 | 432
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 296 | 305 | 601
Parent study (NI-AC301 or NI-AC302) [Count of Participants; unit: Participants]
  NI-AC301 | 150 | 159 | 309
  NI-AC302 | 146 | 146 | 292

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events Ongoing From Parent Study at Start of Study NI-AC303)
Description: This outcome measure shows the number of subjects with at least one ongoing adverse event from the pivotal studies (NI-AC301 and NI-AC302) at the time they rolled over into this study (NI-AC303). The final study visit (Week 12) for the pivotal studies served as the Baseline visit for this study. Subjects who were assigned to SB204 in the pivotal studies are denoted as SB204 Experienced and subjects who were assigned to Vehicle Gel on the pivotal studies are denoted as SB204 Naive.
Time Frame: Baseline
Population: Safety population There were 59 subjects in the SB204 Experienced group with 104 ongoing AEs at the time of rollover and 62 SB204 Naive subjects with 97 ongoing AEs at the time of rollover.
Measure: Count of Participants; unit: Participants
Groups:
- SB204 Experienced: Subjects who were assigned to the SB204 4% QD treatment group in NI-AC301/NI-AC302.
- SB204 Naive: Subjects who were assigned to the Vehicle Gel QD treatment group in NI-AC301/NI-AC302.
Arm/Group | SB204 Experienced | SB204 Naive
Number analyzed (Participants) | 296 | 305
Participants | 59 | 62

2. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events
Description: Number of subjects with adverse events that had an onset date on or after entry into study NI-AC303.
Time Frame: Week 40/End of Treatment
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- SB204 Experienced: Subjects who were assigned to and received SB204 4% QD in the parent (pivotal) study (NI-AC301 or NI-AC302).
- SB204 Naive: Subjects who were assigned to and received Vehicle Gel in the parent (pivotal) study (NI-AC301 or NI-AC302).
Arm/Group | SB204 Experienced | SB204 Naive
Number analyzed (Participants) | 296 | 305
Participants | 54 | 58

3. Secondary Outcome: Tolerability Assessment (Analysis of Tolerability Scores at Each Visit Through End of Treatment)
Description: Analysis of cutaneous tolerability scores at each visit through end of treatment. Baseline is the Week 12 assessment from the previous study (NI-AC301 or NI-AC302). The Cutaneous Tolerability Assessment scale consisted of the investigator's assessment of erythema, scaling, and dryness at the time the assessment was made. Pruritus and burning/stinging were based on the subject's report for the previous 24 hours. Each component was graded on a scale of 0-3, with 0 being none (not present) and 3 being severe. Higher scores indicated a higher severity of reaction.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 36, Week 40
Population: Safety population: per the Statistical Analysis Plan, data are presented for the combined study population of 601 subjects.
Measure: Number; unit: participants
Groups:
- SB204 4%: SB204 4%: Open label, topical SB204 4% once daily.
Arm/Group | SB204 4%
Number analyzed (Participants) | 601
participants
  Baseline: Erythema: none (0): number analyzed (Participants) | 589
  Baseline: Erythema: none (0) | 493
  Baseline: Erythema: mild (1): number analyzed (Participants) | 589
  Baseline: Erythema: mild (1) | 80
  Baseline: Erythema: moderate (2): number analyzed (Participants) | 589
  Baseline: Erythema: moderate (2) | 16
  Baseline: Erythema: severe (3): number analyzed (Participants) | 589
  Baseline: Erythema: severe (3) | 0
  Week 4: Erythema: none (0): number analyzed (Participants) | 584
  Week 4: Erythema: none (0) | 461
  Week 4: Erythema: mild (1): number analyzed (Participants) | 584
  Week 4: Erythema: mild (1) | 109
  Week 4: Erythema: moderate (2): number analyzed (Participants) | 584
  Week 4: Erythema: moderate (2) | 14
  Week 4: Erythema: severe (3): number analyzed (Participants) | 584
  Week 4: Erythema: severe (3) | 0
  Week 12: Erythema: none (0): number analyzed (Participants) | 526
  Week 12: Erythema: none (0) | 432
  Week 12: Erythema: mild (1): number analyzed (Participants) | 526
  Week 12: Erythema: mild (1) | 84
  Week 12: Erythema: moderate (2): number analyzed (Participants) | 526
  Week 12: Erythema: moderate (2) | 10
  Week 12: Erythema: severe (3): number analyzed (Participants) | 526
  Week 12: Erythema: severe (3) | 0
  Week 24: Erythema: none (0): number analyzed (Participants) | 487
  Week 24: Erythema: none (0) | 411
  Week 24: Erythema: mild (1): number analyzed (Participants) | 487
  Week 24: Erythema: mild (1) | 66
  Week 24: Erythema: moderate (2): number analyzed (Participants) | 487
  Week 24: Erythema: moderate (2) | 10
  Week 24: Erythema: severe (3): number analyzed (Participants) | 487
  Week 24: Erythema: severe (3) | 0
  Week 36: Erythema: none (0): number analyzed (Participants) | 450
  Week 36: Erythema: none (0) | 385
  Week 36: Erythema: mild (1): number analyzed (Participants) | 450
  Week 36: Erythema: mild (1) | 60
  Week 36: Erythema: moderate (2): number analyzed (Participants) | 450
  Week 36: Erythema: moderate (2) | 5
  Week 36: Erythema: severe (3): number analyzed (Participants) | 450
  Week 36: Erythema: severe (3) | 0
  Week 40: Erythema: none (0): number analyzed (Participants) | 448
  Week 40: Erythema: none (0) | 387
  Week 40: Erythema: mild (1): number analyzed (Participants) | 448
  Week 40: Erythema: mild (1) | 57
  Week 40: Erythema: moderate (2): number analyzed (Participants) | 448
  Week 40: Erythema: moderate (2) | 4
  Week 40: Erythema: severe (3): number analyzed (Participants) | 448
  Week 40: Erythema: severe (3) | 0
  Week 40/ET: Erythema: none (0): number analyzed (Participants) | 495
  Week 40/ET: Erythema: none (0) | 419
  Week 40/ET Erythema: mild (1): number analyzed (Participants) | 495
  Week 40/ET Erythema: mild (1) | 70
  Week 40/ET: Erythema: moderate (2): number analyzed (Participants) | 495
  Week 40/ET: Erythema: moderate (2) | 6
  Week 40/ET: Erythema: severe (3): number analyzed (Participants) | 495
  Week 40/ET: Erythema: severe (3) | 0
  Baseline: Scaling: none (0): number analyzed (Participants) | 589
  Baseline: Scaling: none (0) | 553
  Baseline: Scaling: mild (1): number analyzed (Participants) | 589
  Baseline: Scaling: mild (1) | 33
  Baseline: Scaling: moderate (2): number analyzed (Participants) | 589
  Baseline: Scaling: moderate (2) | 3
  Baseline: Scaling: severe (3): number analyzed (Participants) | 589
  Baseline: Scaling: severe (3) | 0
  Week 4: Scaling: none (0): number analyzed (Participants) | 584
  Week 4: Scaling: none (0) | 535
  Week 4: Scaling: mild (1): number analyzed (Participants) | 584
  Week 4: Scaling: mild (1) | 46
  Week 4: Scaling: moderate (2): number analyzed (Participants) | 584
  Week 4: Scaling: moderate (2) | 3
  Week 4: Scaling: severe (3): number analyzed (Participants) | 584
  Week 4: Scaling: severe (3) | 0
  Week 12: Scaling: none (0): number analyzed (Participants) | 526
  Week 12: Scaling: none (0) | 487
  Week 12: Scaling: mild (1): number analyzed (Participants) | 526
  Week 12: Scaling: mild (1) | 37
  Week 12: Scaling: moderate (2): number analyzed (Participants) | 526
  Week 12: Scaling: moderate (2) | 2
  Week 12: Scaling: severe (3): number analyzed (Participants) | 526
  Week 12: Scaling: severe (3) | 0
  Week 24: Scaling: none (0): number analyzed (Participants) | 487
  Week 24: Scaling: none (0) | 449
  Week 24: Scaling: mild (1): number analyzed (Participants) | 487
  Week 24: Scaling: mild (1) | 35
  Week 24: Scaling: moderate (2): number analyzed (Participants) | 487
  Week 24: Scaling: moderate (2) | 3
  Week 24: Scaling: severe (3): number analyzed (Participants) | 487
  Week 24: Scaling: severe (3) | 0
  Week 36: Scaling: none (0): number analyzed (Participants) | 450
  Week 36: Scaling: none (0) | 398
  Week 36: Scaling: mild (1): number analyzed (Participants) | 450
  Week 36: Scaling: mild (1) | 51
  Week 36: Scaling: moderate (2): number analyzed (Participants) | 450
  Week 36: Scaling: moderate (2) | 1
  Week 36: Scaling: severe (3): number analyzed (Participants) | 450
  Week 36: Scaling: severe (3) | 0
  Week 40: Scaling: none (0): number analyzed (Participants) | 448
  Week 40: Scaling: none (0) | 423
  Week 40: Scaling: mild (1): number analyzed (Participants) | 448
  Week 40: Scaling: mild (1) | 25
  Week 40: Scaling: moderate (2): number analyzed (Participants) | 448
  Week 40: Scaling: moderate (2) | 0
  Week 40: Scaling: severe (3): number analyzed (Participants) | 448
  Week 40: Scaling: severe (3) | 0
  Week 40/ET: Scaling: none (0): number analyzed (Participants) | 495
  Week 40/ET: Scaling: none (0) | 462
  Week 40/ET: Scaling: mild (1): number analyzed (Participants) | 495
  Week 40/ET: Scaling: mild (1) | 32
  Week 40/ET: Scaling: moderate (2): number analyzed (Participants) | 495
  Week 40/ET: Scaling: moderate (2) | 1
  Week 40/ET: Scaling: severe (3): number analyzed (Participants) | 495
  Week 40/ET: Scaling: severe (3) | 0
  Baseline: Dryness: none (0): number analyzed (Participants) | 589
  Baseline: Dryness: none (0) | 510
  Baseline: Dryness: mild (1): number analyzed (Participants) | 589
  Baseline: Dryness: mild (1) | 73
  Baseline: Dryness: moderate (2): number analyzed (Participants) | 589
  Baseline: Dryness: moderate (2) | 6
  Baseline: Dryness: severe (3): number analyzed (Participants) | 589
  Baseline: Dryness: severe (3) | 0
  Week 4: Dryness: none (0): number analyzed (Participants) | 584
  Week 4: Dryness: none (0) | 496
  Week 4: Dryness: mild (1): number analyzed (Participants) | 584
  Week 4: Dryness: mild (1) | 82
  Week 4: Dryness: moderate (2): number analyzed (Participants) | 584
  Week 4: Dryness: moderate (2) | 6
  Week 4: Dryness: severe (3): number analyzed (Participants) | 584
  Week 4: Dryness: severe (3) | 0
  Week 12: Dryness: none (0): number analyzed (Participants) | 526
  Week 12: Dryness: none (0) | 440
  Week 12: Dryness: mild (1): number analyzed (Participants) | 526
  Week 12: Dryness: mild (1) | 82
  Week 12: Dryness: moderate (2): number analyzed (Participants) | 526
  Week 12: Dryness: moderate (2) | 4
  Week 12: Dryness: severe (3): number analyzed (Participants) | 526
  Week 12: Dryness: severe (3) | 0
  Week 24: Dryness: none (0): number analyzed (Participants) | 487
  Week 24: Dryness: none (0) | 398
  Week 24: Dryness: mild (1): number analyzed (Participants) | 487
  Week 24: Dryness: mild (1) | 80
  Week 24: Dryness: moderate (1): number analyzed (Participants) | 487
  Week 24: Dryness: moderate (1) | 7
  Week 24: Dryness: severe (3): number analyzed (Participants) | 487
  Week 24: Dryness: severe (3) | 2
  Week 36: Dryness: none (0): number analyzed (Participants) | 450
  Week 36: Dryness: none (0) | 382
  Week 36: Dryness: mild (1): number analyzed (Participants) | 450
  Week 36: Dryness: mild (1) | 68
  Week 36: Dryness: moderate (2): number analyzed (Participants) | 450
  Week 36: Dryness: moderate (2) | 0
  Week 36: Dryness: severe (3): number analyzed (Participants) | 450
  Week 36: Dryness: severe (3) | 0
  Week 40: Dryness: none (0): number analyzed (Participants) | 448
  Week 40: Dryness: none (0) | 386
  Week 40: Dryness: mild (1): number analyzed (Participants) | 448
  Week 40: Dryness: mild (1) | 61
  Week 40: Dryness: moderate (2): number analyzed (Participants) | 448
  Week 40: Dryness: moderate (2) | 1
  Week 40: Dryness: severe (3): number analyzed (Participants) | 448
  Week 40: Dryness: severe (3) | 0
  Week 40/ET: Dryness: none (0): number analyzed (Participants) | 495
  Week 40/ET: Dryness: none (0) | 422
  Week 40/ET Dryness: mild (1): number analyzed (Participants) | 495
  Week 40/ET Dryness: mild (1) | 70
  Week 40/ET: Dryness: moderate (2): number analyzed (Participants) | 495
  Week 40/ET: Dryness: moderate (2) | 2
  Week 40/ET Week 40/ET: Dryness: severe (3): number analyzed (Participants) | 495
  Week 40/ET Week 40/ET: Dryness: severe (3) | 1
  Baseline: Pruritus: none (0): number analyzed (Participants) | 589
  Baseline: Pruritus: none (0) | 560
  Baseline: Pruritus: mild (1): number analyzed (Participants) | 589
  Baseline: Pruritus: mild (1) | 26
  Baseline: Pruritus: moderate (2): number analyzed (Participants) | 589
  Baseline: Pruritus: moderate (2) | 3
  Baseline: Pruritus: severe (3) Baseline: Pruritus: severe (3): number analyzed (Participants) | 589
  Baseline: Pruritus: severe (3) Baseline: Pruritus: severe (3) | 0
  Week 4: Pruritus: none (0): number analyzed (Participants) | 584
  Week 4: Pruritus: none (0) | 540
  Week 4: Pruritus: mild (1): number analyzed (Participants) | 584
  Week 4: Pruritus: mild (1) | 40
  Week 4: Pruritus: moderate (2): number analyzed (Participants) | 584
  Week 4: Pruritus: moderate (2) | 2
  Week 4: Pruritus: severe (3): number analyzed (Participants) | 584
  Week 4: Pruritus: severe (3) | 2
  Week 12: Pruritus: none (0): number analyzed (Participants) | 526
  Week 12: Pruritus: none (0) | 481
  Week 12: Pruritus: mild (2): number analyzed (Participants) | 526
  Week 12: Pruritus: mild (2) | 40
  Week 12: Pruritus: moderate (2): number analyzed (Participants) | 526
  Week 12: Pruritus: moderate (2) | 3
  Week 12: Pruritus: severe (3): number analyzed (Participants) | 526
  Week 12: Pruritus: severe (3) | 2
  Week 24: Pruritus: none (0): number analyzed (Participants) | 487
  Week 24: Pruritus: none (0) | 454
  Week 24: Pruritus: Week 24 mild (1): number analyzed (Participants) | 487
  Week 24: Pruritus: Week 24 mild (1) | 30
  Week 24: Pruritus: moderate (2): number analyzed (Participants) | 487
  Week 24: Pruritus: moderate (2) | 2
  Week 24: Pruritus: 24 severe (3): number analyzed (Participants) | 487
  Week 24: Pruritus: 24 severe (3) | 1
  Week 36: Pruritus: none (0): number analyzed (Participants) | 450
  Week 36: Pruritus: none (0) | 429
  Week 36: Pruritus: mild (1): number analyzed (Participants) | 450
  Week 36: Pruritus: mild (1) | 18
  Week 36: Pruritus: moderate (2): number analyzed (Participants) | 450
  Week 36: Pruritus: moderate (2) | 2
  Week 36: Pruritus: severe (3): number analyzed (Participants) | 450
  Week 36: Pruritus: severe (3) | 1
  Week 40: Pruritus: none (0): number analyzed (Participants) | 448
  Week 40: Pruritus: none (0) | 418
  Week 40: Pruritus: mild (1): number analyzed (Participants) | 448
  Week 40: Pruritus: mild (1) | 29
  Week 40: Pruritus: moderate (2): number analyzed (Participants) | 448
  Week 40: Pruritus: moderate (2) | 0
  Week 40: Pruritus: severe (3): number analyzed (Participants) | 448
  Week 40: Pruritus: severe (3) | 1
  Week 40/ET: Pruritus: none (0): number analyzed (Participants) | 495
  Week 40/ET: Pruritus: none (0) | 457
  Week 40/ET: Pruritus: mild (1): number analyzed (Participants) | 495
  Week 40/ET: Pruritus: mild (1) | 34
  Week 40/ET: Pruritus: moderate (2): number analyzed (Participants) | 495
  Week 40/ET: Pruritus: moderate (2) | 0
  Week 40/ET: Pruritus: severe (3): number analyzed (Participants) | 495
  Week 40/ET: Pruritus: severe (3) | 4
  Baseline Burning/Stinging: none (0): number analyzed (Participants) | 589
  Baseline Burning/Stinging: none (0) | 536
  Baseline Burning/Stinging: mild (1): number analyzed (Participants) | 589
  Baseline Burning/Stinging: mild (1) | 53
  Baseline Burning/Stinging: moderate (2): number analyzed (Participants) | 589
  Baseline Burning/Stinging: moderate (2) | 0
  Baseline Burning/Stinging: severe (3): number analyzed (Participants) | 589
  Baseline Burning/Stinging: severe (3) | 0
  Week 4: Burning/Stinging: none (0): number analyzed (Participants) | 584
  Week 4: Burning/Stinging: none (0) | 512
  Week 4: Burning/Stinging: mild (1): number analyzed (Participants) | 584
  Week 4: Burning/Stinging: mild (1) | 65
  Week 4: Burning/Stinging: moderate (2): number analyzed (Participants) | 584
  Week 4: Burning/Stinging: moderate (2) | 7
  Week 4: Burning/Stinging: severe (3): number analyzed (Participants) | 584
  Week 4: Burning/Stinging: severe (3) | 0
  Week 12: Burning/Stinging: none (0): number analyzed (Participants) | 526
  Week 12: Burning/Stinging: none (0) | 463
  Week 12: Burning/Stinging: mild (1): number analyzed (Participants) | 526
  Week 12: Burning/Stinging: mild (1) | 56
  Week 12: Burning/Stinging: moderate (2): number analyzed (Participants) | 526
  Week 12: Burning/Stinging: moderate (2) | 7
  Week 12: Burning/Stinging: severe (3): number analyzed (Participants) | 526
  Week 12: Burning/Stinging: severe (3) | 0
  Week 24: Burning/Stinging: none (0): number analyzed (Participants) | 487
  Week 24: Burning/Stinging: none (0) | 436
  Week 24: Burning/Stinging: mild (1): number analyzed (Participants) | 487
  Week 24: Burning/Stinging: mild (1) | 50
  Week 24: Burning/Stinging: moderate (2): number analyzed (Participants) | 487
  Week 24: Burning/Stinging: moderate (2) | 1
  Week 24: Burning/Stinging: severe (3): number analyzed (Participants) | 487
  Week 24: Burning/Stinging: severe (3) | 0
  Week 36: Burning/Stinging: none (0): number analyzed (Participants) | 450
  Week 36: Burning/Stinging: none (0) | 422
  Week 36: Burning/Stinging: mild (1): number analyzed (Participants) | 450
  Week 36: Burning/Stinging: mild (1) | 25
  Week 36: Burning/Stinging: moderate (2): number analyzed (Participants) | 450
  Week 36: Burning/Stinging: moderate (2) | 3
  Week 36: Burning/Stinging: severe (3): number analyzed (Participants) | 450
  Week 36: Burning/Stinging: severe (3) | 0
  Week 40: Burning/Stinging: none (0): number analyzed (Participants) | 448
  Week 40: Burning/Stinging: none (0) | 411
  Week 40: Burning/Stinging: mild: number analyzed (Participants) | 448
  Week 40: Burning/Stinging: mild | 36
  Week 40: Burning/Stinging: moderate (2): number analyzed (Participants) | 448
  Week 40: Burning/Stinging: moderate (2) | 1
  Week 40: Burning/Stinging: severe (3): number analyzed (Participants) | 448
  Week 40: Burning/Stinging: severe (3) | 0
  Week 40/ET: Burning/Stinging: none (0): number analyzed (Participants) | 495
  Week 40/ET: Burning/Stinging: none (0) | 451
  Week 40/ET: Burning/Stinging: mild (1): number analyzed (Participants) | 495
  Week 40/ET: Burning/Stinging: mild (1) | 40
  Week 40/ET: Burning/Stinging: moderate (2): number analyzed (Participants) | 495
  Week 40/ET: Burning/Stinging: moderate (2) | 2
  Week 40/ET: Burning/Stinging: severe (3): number analyzed (Participants) | 495
  Week 40/ET: Burning/Stinging: severe (3) | 2

4. Secondary Outcome: Inflammatory Lesion Counts by Study Visit
Description: Absolute count of inflammatory lesions at each visit (face only)--safety population
Time Frame: Baseline through Week 40
Population: Safety population
Measure: Mean (Standard Deviation); unit: number of inflammatory lesions
Groups:
- SB204 4% Experienced: Subjects who received SB204 % QD in the parent trial (NI-AC301 or NI-AC302)
- SB204 Naive: Subjects who received vehicle gel in the parent trial (NI-AC301 or NI-AC302) and received SB204 4% QD in this trial.
Arm/Group | SB204 4% Experienced | SB204 Naive
Number analyzed (Participants) | 296 | 305
number of inflammatory lesions
  Baseline: number analyzed (Participants) | 293 | 296
  Baseline | 13.2 (9.94) | 15.3 (10.81)
  Week 4: number analyzed (Participants) | 291 | 293
  Week 4 | 12.2 (9.98) | 14.3 (10.27)
  Week 12: number analyzed (Participants) | 268 | 258
  Week 12 | 10.8 (9.66) | 13.1 (9.74)
  Week 24: number analyzed (Participants) | 254 | 233
  Week 24 | 10.3 (7.5) | 11.4 (9.41)
  Week 36: number analyzed (Participants) | 235 | 215
  Week 36 | 8.3 (8.39) | 9.7 (9.11)
  Week 40: number analyzed (Participants) | 232 | 216
  Week 40 | 7.3 (8.13) | 8.9 (8.99)
  Week 40/ET: number analyzed (Participants) | 249 | 246
  Week 40/ET | 7.9 (8.47) | 9.8 (9.46)

5. Secondary Outcome: Non-Inflammatory Lesion Counts by Study Visit
Description: Absolute count of non-inflammatory lesions by study visit (face only)
Time Frame: Baseline through Week 40
Population: Safety population
Measure: Mean (Standard Deviation); unit: number of non-inflammatory lesions
Groups:
- SB204 4% Experienced: Subjects who received SB204 4% in the parent study.
- SB204 Naive: Subjects who received vehicle gel in the parent study and SB204 4% in this open label study.
Arm/Group | SB204 4% Experienced | SB204 Naive
Number analyzed (Participants) | 296 | 305
number of non-inflammatory lesions
  Baseline: number analyzed (Participants) | 293 | 296
  Baseline | 23.6 (16.08) | 25.5 (18.32)
  Week 4: number analyzed (Participants) | 291 | 293
  Week 4 | 21.9 (16.27) | 23.0 (16.07)
  Week 12: number analyzed (Participants) | 268 | 258
  Week 12 | 19.7 (15.14) | 21.5 (16.09)
  Week 24: number analyzed (Participants) | 254 | 233
  Week 24 | 17.2 (14.67) | 17.5 (13.20)
  Week 36: number analyzed (Participants) | 235 | 215
  Week 36 | 14.0 (13.19) | 15.4 (13.06)
  Week 40: number analyzed (Participants) | 232 | 216
  Week 40 | 12.6 (13.77) | 14.1 (12.59)
  Week 40/ET: number analyzed (Participants) | 249 | 246
  Week 40/ET | 13.7 (14.64) | 15.4 (14.70)

ADVERSE EVENTS:
Time Frame: Baseline through Week 40 (approximately 9 months)
Description: Treatment emergent adverse events (TEAEs) were defined as AEs reported on or after the first day of enrollment in this long term safety study. They are reported for the combined study safety population (SB204 experienced + SB204 naive).
Groups:
- SB204 Experienced: Subjects who received SB204 4% QD in the parent study (NI-AC301 or NI-AC302) and continued to receive open label SB204 4% QD in this study.
- SB204 Naive: Subjects who received vehicle gel QD in the parent study (NI-AC301 or NI-AC302) and SB204 4% QD in this study.
Arm/Group | SB204 Experienced | SB204 Naive
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/305
Serious Adverse Events (participants affected / at risk) | 4/296 | 2/305
Other Adverse Events (participants affected / at risk) | 34/296 | 32/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB204 Experienced (N=296) | SB204 Naive (N=305)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Conduct Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB204 Experienced (N=296) | SB204 Naive (N=305)
Nasopharyngitis (Infections and infestations) | 5 | 14
Influenza (Infections and infestations) | 4 | 3
Application site dryness (General disorders) | 8 | 3
Application site pruritus (General disorders) | 3 | 6
Application site pain (General disorders) | 3 | 4
Headache (Nervous system disorders) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02798120/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT02798120/SAP_001.pdf